CLINICAL TRIAL: NCT01250613
Title: Genomic Study of Congenital Malformation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: Academia Sinica, Taiwan (Other)
Responsible Party: Fuu-Jen Tsai, China Medical University Hospital
Other Study IDs: DMR99-IRB-037
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Genomic Aberrations in Patients Diagnosed as Congenital Malformation With Unknown Etiology

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Genomic aberrations in patients diagnosed as congenital malformation with unknown etiology will be identified using high-density oligonucleotide array.

DETAILED DESCRIPTION:
The Affymetrix GeneChip® Human Mapping SNP 6.0 array, includes more than 900,000 SNP probes plus more than 900,000 CNV probes in a single chip, can provide high density makers information for the human genome. The median inter-marker distance is 670 bases and the average inter-marker distance is 1.67 kb, and the resolution can be as high as 200 kb. The Affymetrix® Cytogenetics Whole-Genome 2.7M Array gives the greatest power to detect known and novel chromosome aberrations across the entire genome. In addition, the whole-genome array includes 400,000 single nucleotide polymorphisms (SNPs) to enable the detection of loss of heterozygosity (LOH), uniparental disomy (UPD), and regions identical-by-descent.

If we are able to identify the candidate genomic regions that are associated with the congenital malformation/syndrome, we may have a better chance to understand the pathogenesis of congenital malformation/syndrome as well as the mechanisms underlying the abnormal chromosome rare diseases. The results from this study can also facilitate the clinical diagnosis and provide genetic basis for consultation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is diagnosed as congenital malformation/syndromes.
2. Participants can be any ages, and both males and females are eligible.
3. Subjects agree and are capable of giving informed consent. If participants are under 18 years old or incapable of giving consent, an informed consent must be approved by their legal guardians.
4. Availability and willingness of the proband and first-degree biological family (parents, full sibling, or adult-age offspring) who also meets the same congenital malformation syndrome.
5. Availability and willingness of the proband's biological parents whatever with or without the same congenital malformation syndrome.

Exclusion Criteria:

1. Subject or legal guardian is unable to understand or give informed consent.
2. The molecular cause for congenital malformation/syndromes of subjects or their affected first-degree biological family (parents, full sibling, or adult-age offspring) can be revealed by karyotype assay or FISH.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Genomic aberrations in patients diagnosed as congenital malformation with unknown etiology
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2010-06

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan